CLINICAL TRIAL: NCT01480739
Title: A Randomised, Double-blind, Placebo-Controlled, Two-way Cross-over, Single Centre Study in Healthy Subjects to Assess the Effect of Oral Dosing of AZD5069 on Neutrophil Number and Function in Peripheral Blood and the Ability to Recruit Neutrophils Into the Circulation After Exercise and Subcutaneous
Brief Title: AZD5069 Neutrophil Function Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D3550C00017
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Chemokine Receptor 2 (CXCR2) Antagonist
Keywords: Phase 1, AZD5069, safety and tolerability, healthy volunteer,
MeSH Terms: interventions — N-(2-(2,3-difluoro-6-benzylthio)-6-(3,4-dihydroxybutan-2-yloxy)pyrimidin-4-yl)azetidine-1-sulfonamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): AZD5069 100 mg capsules (50 mg BD) for 7 days
  Interventions: Drug: 100 mg (50 mg x 2) AZD5069
- 2 (Experimental): Placebo twice daily for 7 days
  Interventions: Drug: 100 mg Placebo

INTERVENTIONS:
Drug: 100 mg (50 mg x 2) AZD5069 — Twice daily for 7 days
  Arms: 1
Drug: 100 mg Placebo — Twice daily for 7 days
  Arms: 2

SUMMARY:
Study in healthy volunteer to see effect of AZD5069 and placebo on neutrophil number and function (phagocytosis and oxidative burst) in the circulation, following a burst of strenuous exercise and following subcutaneous injection of granulocyte-colony stimulating factor (G-CSF)

DETAILED DESCRIPTION:
A Randomised, Double-blind, Placebo-Controlled, Two-way Cross-over, Single Centre Study in Healthy Subjects to Assess the Effect of Oral Dosing of AZD5069 on Neutrophil Number and Function in Peripheral Blood and the Ability to Recruit Neutrophils into the Circulation after Exercise and Subcutaneous

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male or post-menopausal/surgical sterile females, aged 18 to 45 years inclusive at screening
* Only women of non-childbearing potential are included in the study, ie, women who are permanently or surgically sterilised or post-menopausal
* Non-smokers or ex-smokers with no smoking history the last 12 months prior to Visit 1 and a smoking history of less than 10 pack years (1 pack year = tobacco consumption corresponding to 20 cigarettes smoked per day for 1 year) at screening
* Body mass index (BMI) >18 kg/m2 and ≤30 kg/m2 and a minimum weight of 50 kg

Exclusion Criteria:

* Subjects with a history of or active or latent tuberculosis (TB), or close contact with anybody with active TB
* Subjects with a history of malignancy or neoplastic disease (except successfully treated basal or squamous cell carcinoma of the skin)
* Subjects who are pyrexial with a body temperature of greater than 37.7 C at Visit 2, or as judged by the Investigator
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) level ≥1.5 x upper limit of normal (ULN) at screening (Visit 2)
* Peripheral blood neutrophils above or below the laboratory reference range at screening (Visit 2) hsCRP above the upper limit of the laboratory reference range at Visit 2

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in status of Neutrophil function (phagocytosis and oxidative burst) in subjects on AZD5069 and placebo | Day -1, Day 1, Day 2, Day 3, Day 4 and 7 days after end of treatment.
Circulating neutrophils during exercise challenge measured by average neutrophil values over time | Pre-dose, 10 min, 2h, 4 hours post exercise test
Circulating neutrophils following subcutaneous injection of granulocyte-colony stimulating factor (G-CSF) | Pre-dose, 2h, 6h, 12h, 24h, 36 hours post subcutaneous G-CSF

SECONDARY OUTCOMES:
Adverse events | Screening to Day 63
Steady state 24 hour pharmacokinetic profile of the AZD5069 capsule following twice daily (bid) dosing | Pre-dose on Days 1 - 4 On Day 3 with sampling pre-dose and at 1h, 2h, 3h, 5h, 8h, and 12 hours post dose
Steady state 24 hour profile of circulating neutrophils following twice daily dosing of AZD5069 and its relationship to plasma concentration | Pre-dose and 1, 2, 3, 5, 8, 12 hours post each dose on Days 1 - 4, Day 6 and Day 7
Changes in baseline of vital signs (blood pressure and pulse), clinical laboratory tests, ECGs, and physical examination findings will be presented | Screening to Day 63

CONTACTS AND LOCATIONS:
Overall Officials: Tim Mant, MD, Principal Investigator — Quintiles research Unit; Bengt Larsson, MD, Study Director — AstraZeneca Medical Science Director
Locations (1):
- London, UK, United Kingdom

REFERENCES:
- [Derived] Cullberg M, Arfvidsson C, Larsson B, Malmgren A, Mitchell P, Wahlby Hamren U, Wray H. Pharmacokinetics of the Oral Selective CXCR2 Antagonist AZD5069: A Summary of Eight Phase I Studies in Healthy Volunteers. Drugs R D. 2018 Jun;18(2):149-159. doi: 10.1007/s40268-018-0236-x. PMID 29856004
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1341&filename=D3550C00017_Study_Synopsis.pdf